CLINICAL TRIAL: NCT01785277
Title: Validation of a Translation Into Spanish (Mexico) of the Spinal Cord Independence Measure III
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Adriana Ivonne Cervantes Vázquez., Chief of the Rehabilitation Department, American British Cowdray Medical Center
Other Study IDs: ABC-SCIM-01-2013
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Independence Measure; SCIM; Spinal cord injury; Traumatic spine injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCIM scores for patients with SCI: All patients with SCI included in the study

SUMMARY:
The propose of the study is to validate in Mexico a spanish translation of the Spinal Cord Independence Measure (SCIM) Version III, in patients with spinal cord injury (SCI).

Internal consistency, reproducibility and reliability will be addressed scoring the results of the translated version at two time frames and also of the same patients by different examiners (physicians, nurses and technicians).

DETAILED DESCRIPTION:
The worldwide estimated annual incidence of SCI has a broad spectrum, ranging from 236 to 1009 cases per million of people. In Mexico there is an estimate of 18.1 cases per million people, affecting primary men in their productive age (25-34 years old).

Most of the patients have disabilities after the injury, and become dependent of their families or professional care providers. The cornerstone treatment in the long therm is rehabilitation and the main goal is to achieve patient independence.

Over the last two decades many disability measure instruments have been developed, like the Functional Interdisciplinary Measure (FIM). This scale though it is very useful for patients' general outcome, it does not grade patients' independence entirely. In 1997, Dr. Amiram Catz developed the first version of the Spinal Cord Independence Measure (SCIM). Since its first version, it showed to be a very powerful tool to assess patients' independence. Recently, the SCIM-III has been validated in a multicenter study, showing validity, reliability and internal consistency.

The aim of this study is to perform a translate and trans-cultural adaptation of the SCIM-III into Spanish and to perform also its validation in Mexican population.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury

Exclusion Criteria:

* Patient with any other injury/lesion that produces dependence or disability

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spinal cord injury.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Patient's change in independence measured by the translated SCIM-III version | Initial evaluation and 7 days after.
  The objective of this outcome is to evaluate the ability of the translated SCIM-III version to asses the patients grade of independence in two different time frames and by two different examiners.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Ivonne Cervantes Vasquez, MD, Principal Investigator — Centro Medico ABC
Locations (1):
- ABC Medical Center, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Cripps RA, Lee BB, Wing P, Weerts E, Mackay J, Brown D. A global map for traumatic spinal cord injury epidemiology: towards a living data repository for injury prevention. Spinal Cord. 2011 Apr;49(4):493-501. doi: 10.1038/sc.2010.146. Epub 2010 Nov 23. PMID 21102572
- [Background] Ho CH, Wuermser LA, Priebe MM, Chiodo AE, Scelza WM, Kirshblum SC. Spinal cord injury medicine. 1. Epidemiology and classification. Arch Phys Med Rehabil. 2007 Mar;88(3 Suppl 1):S49-54. doi: 10.1016/j.apmr.2006.12.001. PMID 17321849
- [Background] Wyndaele M, Wyndaele JJ. Incidence, prevalence and epidemiology of spinal cord injury: what learns a worldwide literature survey? Spinal Cord. 2006 Sep;44(9):523-9. doi: 10.1038/sj.sc.3101893. Epub 2006 Jan 3. PMID 16389270
- [Background] Kirshblum SC, Priebe MM, Ho CH, Scelza WM, Chiodo AE, Wuermser LA. Spinal cord injury medicine. 3. Rehabilitation phase after acute spinal cord injury. Arch Phys Med Rehabil. 2007 Mar;88(3 Suppl 1):S62-70. doi: 10.1016/j.apmr.2006.12.003. PMID 17321851
- [Background] Catz A, Itzkovich M, Agranov E, Ring H, Tamir A. The spinal cord independence measure (SCIM): sensitivity to functional changes in subgroups of spinal cord lesion patients. Spinal Cord. 2001 Feb;39(2):97-100. doi: 10.1038/sj.sc.3101118. PMID 11402366
- [Background] Catz A, Itzkovich M, Agranov E, Ring H, Tamir A. SCIM--spinal cord independence measure: a new disability scale for patients with spinal cord lesions. Spinal Cord. 1997 Dec;35(12):850-6. doi: 10.1038/sj.sc.3100504. PMID 9429264
- [Background] Bluvshtein V, Front L, Itzkovich M, Aidinoff E, Gelernter I, Hart J, Biering-Soerensen F, Weeks C, Laramee MT, Craven C, Hitzig SL, Glaser E, Zeilig G, Aito S, Scivoletto G, Mecci M, Chadwick RJ, El Masry WS, Osman A, Glass CA, Silva P, Soni BM, Gardner BP, Savic G, Bergstrom EM, Catz A. SCIM III is reliable and valid in a separate analysis for traumatic spinal cord lesions. Spinal Cord. 2011 Feb;49(2):292-6. doi: 10.1038/sc.2010.111. Epub 2010 Sep 7. PMID 20820178